CLINICAL TRIAL: NCT06051136
Title: Feasibility of an Early Versus Delayed Rehabilitation Intervention in Patients With Lung Cancer on Cancer-related Fatigue: a Pilot RCT
Brief Title: Early Versus Delayed Rehabilitation Intervention in Patients With Lung Cancer
Acronym: OVER-CRF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: OVER-CRF
Record Dates: First submitted 2023-09-17; First posted 2023-09-22 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Single-center, two-arm, open-label pilot RCT.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The randomization will be done online directly from Smarty, the software that will manage the eCRF for collecting of the study data.
  Furthermore, outcomes will be assessed blindly by staff involved in the research project who do not directly deliver the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early pulmonary rehabilitation (RP) (Experimental): RP immediately after enrollment.
  Interventions: Behavioral: Pulmonary rehabilitation
- Delayed pulmonary rehabilitation (RP) (Experimental): RP after 3 months after enrollment.
  Interventions: Behavioral: Pulmonary rehabilitation

INTERVENTIONS:
Behavioral: Pulmonary rehabilitation — The RP intervention consists in 8 sessions supervised by the physiotherapist weekly or biweekly and 2 therapeutic education group meetings on the importance of exercise and CRF management, over the 3 months of intervention. The RP comprise exercise program performed autonomously at home. Both the outpatient and the autonomously home-based exercise sessions comprise aerobic, resistance and respiratory exercise.
  The exercise program is individualized and can be delivered in telerehabilitation.

SUMMARY:
In Italy, the incidence of lung cancer for the year 2020 has been estimated at about 41.000 new diagnoses. Patients with lung cancer experience debilitating symptoms caused by the disease itself and cancer treatments, such as dyspnea and fatigue, which reduce physical function and quality of life (QoL). It is estimated that 90% of patients undergoing chemotherapy and 57% of patients undergoing lung resection suffer of Cancer-Related Fatigue (CRF).

Previous studies have shown that educational interventions and aerobic and resistance exercise are effective in improving CRF and QoL in patients with lung cancer. However, to date the optimal dose, mode and timing to deliver the intervention during the care pathway for lung cancer patients is unknown. Tolerability and frequency of cancer treatment could be a barrier to adherence to the intervention. Therefore, this study aims to evaluate the feasibility of a rehabilitation intervention aimed at improving CRF with respect to timing of delivery: early vs delayed rehabilitation in lung cancer patients.

DETAILED DESCRIPTION:
The primary outcome of the study is to evaluate the feasibility of the experimental pulmonary rehabilitation (RP) program combining the exercise component with the educational component for patients with lung cancer undergoing chemotherapy and/or radiotherapy and/or immunotherapy, delivering RP at different points in the course of their care pathway. The secondary outcome is to evaluate the impact of the intervention on several health outcomes (CRF, physical performance, and QoL) by assessing any differences between early and delayed RP.

The early RP intervention will be delivered in the first three months of cancer treatment, while the same delayed RP intervention will be delivered three months after the start of treatment. Finally, considering the potential beneficial role that exercise on survival of patients with cancer, this study also aims to evaluate this outcome at 12 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed of stage II and III lung cancer (NSCLC) candidates for anticancer therapies (chemotherapy, radiotherapy, immunotherapy, or combinations thereof), associated or not with surgery. In the last case, patients will be included at least 30 days after surgery.
* Prognosis ≥ 12 months
* At least 18 years old
* Recruited from the pneumology, oncology, radiotherapy, and physical medicine and rehabilitation unit of the Azienda Unità Sanitaria Locale - IRCCS of Reggio Emilia
* Willing and able to give written informed consent

Exclusion Criteria:

* Clinical disorders that contraindicate participation in a moderate exercise program (e.g. preexisting severe physical disabilities, major cognitive or sensory deficits, severe psychiatric disorders, language barrier, etc.).
* NSCLC stage IV
* Patients who are candidates for surgery alone
* Patients who are candidates for neoadjuvant therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-28 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility - Adherence rate to the outpatient RP sessions | At 3 and 6 months after baseline
  The number of patients adhering to at least 70% of outpatient RP sessions scheduled for the relative allocation group will be recorded.

SECONDARY OUTCOMES:
Recruitment rate | At baseline
  The recruitment rate will be estimated with the sample rate calculated as the ratio of the number of patients who partecipate to the study to the number of patients to whom the study is proposed.
Dropout rate | At 3 and 6 months after baseline
  Number of treatment failures, their causes, and number of sessions conducted
Cancer-related fatigue (CRF) | At baseline, at 3, 6, and 12 months after baseline
  CRF will be measured with The Functional Assessment of Chronic Illness Therapy - Fatigue Scale (FACIT-F). The score ranges from 0 to 52. Higher score represents less fatigue experienced by patient. The minimum clinically significant difference for the FACIT-F scale has been estimated at 3 points.
Quality of life (QoL) | At baseline, at 3, 6, and 12 months after baseline
  QoL will be measured by EORTC- QLQ-C30 questionnaire. The QLQ-C30 consists of 30 items, which assess various dimensions of HRQL: five scales of functioning (physical, role, emotional, cognitive and social), three scales assessing symptoms (fatigue, pain and nausea) and a global measure of health status. The remaining six single-question scales assess symptoms: dyspnea, loss of appetite, sleep disorders, constipation and diarrhea, and the perceived economic impact of treating the disease. High scores indicate better HRQL for global health status and functioning scales, but worse symptoms. The minimum clinically significant difference for the EORTC QLQ-C30 scale was estimated to be between 5 and 10 points.
Physical performance | At baseline, at 3 and 6 months after baseline
  Physical performance will be neasured by six minute walk test (6MWT). The 6MWT consists of measuring the distance covered in six minutes. Saturation, heart rate, respiratory and muscle fatigue and the number of stops are also releved at both the start and finish. The minimum clinically significant difference for the 6MWT in lung cancer patients was estimated to be 42 m.
Adherence to the exercise home-based sessions | At baseline, at 3 and 6 months after baseline
  Number of exercise home-based sessions performed by each patient
Physical activity level | At baseline, at 3, 6, and 12 months after baseline
  Physical activity level will be measured by the International Physical Activity Questionnaire - Short Form (IPAQ-SF). IPAQ-SF is a questionnaire used to estimate the amount of physical activity during the previous 7 days. Weekly frequency and average duration of vigorous and moderate physical activity and walking (regardless of whether during work or leisure time) and the number of daily hours spent sitting are asked. In addition, to assess the level of physical activity performed, IPAQ uses METs (Metabolic Equivalent Tasks).
Adverse events | At 3, 6, and 12 months after baseline
  Recording of adverse events related to the exercise intervention during the 6-month intervention period (falls, fractures, muscle pain, exertional dyspnea, acute inflammation of joints stressed in the rehabilitation program, hematomas, etc.).
Survival | At 12 months after baseline

CONTACTS AND LOCATIONS:
Overall Officials: Stefania Fugazzaro, Dr., Principal Investigator — Azienda USL Reggio Emilia - IRCCS
Locations (1):
- Azienda Unità Sanitaria Locale - IRCCS di Reggio Emilia, Reggio Emilia, Reggio Emilia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fugazzaro S, Mainini C, Pecorari A, Denti M, Galavotti MB, Messori M, Costi S, Ciammella P, Falco F, Zanelli F, Cavuto S, Bressi B. Feasibility of an early versus delayed rehabilitation intervention in patients with lung cancer on cancer-related fatigue: a pilot RCT. Future Oncol. 2026 Jan;22(2):147-156. doi: 10.1080/14796694.2025.2607632. Epub 2026 Jan 6. PMID 41496492